CLINICAL TRIAL: NCT03169751
Title: An Exploratory Trial Using sEMG to Differentiate PNES From Epileptic Seizures
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brain Sentinel (Other)
Responsible Party: Sponsor
Other Study IDs: PNES-1.5-11.2016-EU
Record Dates: First submitted 2017-04-20; First posted 2017-05-30 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Non-Epileptic Seizure; Motor Seizure; Epilepsy
MeSH Terms: conditions — Seizures; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- PNES Cohort: Participants who experience a non-epileptic event with upper extremity motor involvement, while enrolled in the trial
  Interventions: Device: Brain Sentinel Monitoring and Alerting System
- Epileptic Cohort: Participants who experience an epileptic event with upper extremity motor involvement, while enrolled in the trial
  Interventions: Device: Brain Sentinel Monitoring and Alerting System

INTERVENTIONS:
Device: Brain Sentinel Monitoring and Alerting System — The Brain Sentinel Monitoring and Alerting System is indicated for use as an adjunct to seizure monitoring in adults in the home or healthcare facilities during periods of rest. The device is to be used on the belly of the biceps muscle to analyze surface electromyographs (sEMG) signals that may be associated with generalized tonic-clonic (GTC) seizures and to provide an alarm to alert caregivers of unilateral, appendicular, tonic extension that could be associated with a GTC seizure. The System records and stores sEMG data for subsequent review by a trained healthcare professional.

SUMMARY:
This is an observational study of subjects receiving standard of care therapy, while admitted to Epilepsy Monitoring Unit, Department of Neurology, General Hospital Hietzing with Neurological Center Rosenhügel. Additional monitoring provided by the SPEAC System will be compared to the gold standard, vEEG. The SPEAC System is being evaluated while being used in adjunct to standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a suspected history of PNES with upper extremity motor involvement or epileptic seizures with upper extremity motor involvement.
2. Is being admitted to a hospital for routine vEEG monitoring related to seizures.
3. Male or female between the ages of 18-99.
4. If female and of childbearing potential, has a negative pregnancy test.
5. Can understand and sign written informed consent prior to the performance of any study assessments.
6. Subject must be competent to follow all study procedures.

Exclusion Criteria:

1.Intracranial EEG electrodes are being used.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with a suspected history of Psychogenic Non Epileptic Seizures with upper extremity motor involvement. and/or Epileptic Seizures with upper extremity motor involvement
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
3 independent physicians' abilities to differentiate between epileptic events (with upper extremity motor involvement) and PNES (with upper extremity motor involvement) using vEEG, using a majority rules approach (2 out of 3) | 5 days
  The primary endpoint is to test a physician's ability to differentiate between epileptic events (with upper extremity motor involvement) and PNES (with upper extremity motor involvement) using vEEG review. PNES and epileptic seizures will initially be identified, described, and documented following routine clinical care (vEEG).
3 independent physicians' abilities to differentiate between epileptic events (with upper extremity motor involvement) and PNES (with upper extremity motor involvement) using sEMG, using a majority rules approach (2 out of 3) | 5 days
  The primary endpoint is to test a physician's ability to differentiate between epileptic events (with upper extremity motor involvement) and PNES (with upper extremity motor involvement) using sEMG recorded by the SPEAC System. PNES and epileptic seizures will initially be identified, described, and documented following routine clinical care (vEEG). The sEMG record will be evaluated to identify PNES, displaying upper extremity motor components, and epileptic seizures, displaying upper extremity (UE) motor components. It is anticipated that > 70% of PNES with UE motor involvement identified by vEEG will be identified by sEMG recordings as well.

SECONDARY OUTCOMES:
To evaluate the System's ability to detect GTC seizures, as compared to vEEG monitoring | 5 days
  It is anticipated that >70% of GTC seizures identified by vEEG will be identified by the SPEAC System's automated alarms as well.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Baumgartner, MD, Principal Investigator — Krankenhaus Hietzing mit Neurologischem Zentrum Rosenhügel
Locations (1):
- Krankenhaus Hietzing mit Neurologischem Zentrum Rosenhugel, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No